CLINICAL TRIAL: NCT01866657
Title: NIRS-Based Cerebral Oximetry Monitoring in Elderly Thoracic Surgical Patients Undergoing Single Lung Ventilation Procedures: A Single Center, Prospective, Randomized Controlled Pilot Study Assessing the Clinical Impact of NIRS-Guided Intervention
Brief Title: Cerebral Oximetry in Single Lung Ventilation Thoracic Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UHCMC-CEROX-01
Record Dates: First submitted 2013-05-12; First posted 2013-05-31 (Estimated); Results first posted 2022-07-05 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-07

CONDITIONS: Hypoxia
Keywords: cerebral oximetry; randomized controlled pilot study; thoracic surgery; single lung ventilation
MeSH Terms: conditions — Hypoxia | interventions — Vasoconstrictor Agents; Phenylephrine; Ephedrine; Dopamine; Sevoflurane; Propofol

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention cohort (Experimental): Open cerebral oximetry monitoring; observed desaturations will be treated with an intervention algorithm including increase FiO2, head/neck repositioning,vasoconstrictor agents, IV fluid bolus, increase ETCO2, additional anesthesia, RBC transfusion.
  Interventions: Drug: Vasoconstrictor Agents; Other: Head/neck repositioning; Other: Increase ETCO2; Other: IV fluid bolus; Drug: Additional anesthesia; Biological: RBC transfusion; Drug: Increase FiO2
- Blinded cerebral oximetry monitoring (No Intervention): These subjects will have continous cerebral oximetry monitoring like the experimental cohort but the values will be blinded to all clinicians and research staff. There will be no cerebral desaturation interventions in this group because the clinicians will not be aware of a desaturation as the monitor's output is blinded in this group.

INTERVENTIONS:
Drug: Vasoconstrictor Agents — cerebral desaturations may be treated with IV vasoactives to increase blood pressure or cardiac output at attending physician's descretion.
  Other Names: phenylephrine, ephedrine, dopamine
  Arms: Intervention cohort
Other: Head/neck repositioning — Assure that arterial and venous neck blood flow is not obstructed related to patient positioning
  Other Names: neck repositioning
  Arms: Intervention cohort
Other: Increase ETCO2 — Allow normalization or slight increase in end tidal CO2 to cause selective cerebral vasodilation and increased tissue blood flow/O2 delivery
  Other Names: Normalize end tidal CO2
  Arms: Intervention cohort
Other: IV fluid bolus — Administer IV fluids to increase preload and cardiac output
  Arms: Intervention cohort
Drug: Additional anesthesia — By deepening anesthetic there will be a decrease in cerebral metabolic oxygen consumption.
  Other Names: sevoflurane, propofol
  Arms: Intervention cohort
Biological: RBC transfusion — By administering RBCs there will be a increase in intravascular volume and cardiac preload and an increase in oxygen carrying capacity
  Arms: Intervention cohort
Drug: Increase FiO2 — Increase FiO2 to improve oxygen delivery to tissue
  Other Names: Increase fractional concentration of inspired oxygen
  Arms: Intervention cohort

SUMMARY:
This is a prospective, randomized controlled pilot study of cerebral oximetry use in elderly patients undergoing thoracic surgical procedures that require the use of single lung ventilation. The hypothesis is that subjects randomized to open cerebral oximetry monitoring that have active intervention to mitigate observed desaturations will have measurable postoperative clinical outcome benefits when compared to the patients randomized to blinded cerebral oximetry monitoring with no active interventions to mitigate desaturations.

DETAILED DESCRIPTION:
Study Rationale The use of bi-frontal, near infrared spectrophotometry (NIRS) based cerebral oximetry monitoring has been demonstrated to result in improved clinical outcomes in both general surgery patients and cardiac surgical patients using prospective, randomized controlled trial methodology. Elderly thoracic surgical patients undergoing procedures that involve single lung ventilation may also stand to benefit from the application of intraoperative and early postoperative NIRS cerebral oximetry monitoring. Cerebral oximetry has not been established as a standard of care monitoring modality in this patient population, thus permitting the application of randomized, controlled testing methodology to assess the potential impact of this monitoring modality upon these patients.

Hypothesis and Objectives:

The primary hypothesis in this pilot study of elderly thoracic surgical patients undergoing procedures involving single lung ventilation (SLV) is that there will be a measurable and significant clinical benefit (as assessed by a broad range of postoperative clinical outcome measures) to the subjects randomized to the intervention cohort (open bi-frontal NIRS based cerebral oximetry monitoring with a standardized intervention protocol) vs. the control cohort (blinded bi-frontal NIRS based cerebral oximetry monitoring).

The primary objective of this pilot study is to identify the most relevant clinical outcome variables which significantly diverge as a result of being randomized to the intervention cohort vs. the control cohort so that a larger, multicenter, prospective, randomized controlled clinical trial can be designed to further test the primary hypothesis as stated in the preceding section. The subsequent larger, multicenter trial will be conducted to definitively demonstrate the ability of INVOS® 5100 guided NIRS-based bi-frontal monitoring to improve clinical outcomes in this surgical patient group and potentially establish a new U.S. Food and Drug Administration cleared indication for this monitoring modality. The clinical outcome variables being assessed as the primary objective are many and a detailed list of these variables can be found in the OUTCOME MEASURES - Primary Outcome Measure Section of this submission.

Secondary objectives of this pilot study include the following:

1. Assess the frequency of cerebral desaturations in both the intervention and control cohorts by examining both the total number of patients experiencing any cerebral desaturation as well as the total number of events among patients experiencing any cerebral desaturation (of at least 5% below baseline and progressively larger desaturations). These analyses will be conducted on the entire study population as well as upon each cohort. The Area Under the Curve (AUC) analysis technique [incremental desaturation categories will be assessed based upon 5 to 50% decreases, measured in 5% increments, from established room air pre-incision baseline as well as oxygen supplemented pre-incision baseline as well as desaturations below absolute measured rSO2 values] will be employed to conduct these analyses.
2. Assess the frequency of adverse clinical events and serious adverse events overall and in each cohort.
3. Perform a comprehensive assessment of the frequency and efficacy of predefined rSO2 desaturation mitigation interventions and their collective ability to affect the observed cerebral oximetry values.
4. Assess the interventional cohort's preoperative demographics and collected covariates for association with the ease or difficulty of mitigating observed cerebral desaturation events.

Exploratory analyses will include performing all possible comparisons of the two groups based upon all collected perioperative variables to examine the potentially significant relationships between the collected clinical variables representing surrogates of organ perfusion/function and cerebral oximetry desaturations (AUCrSO2). The following exploratory endpoints will be assessed:

1. Logistic regression analysis to determine the most relevant AUCrSO2 desaturation value(s) associated with any detrimental clinical outcome(s) monitored in this study
2. Logistic regression analysis to determine the most relevant AUC blood pressure values associated with any detrimental clinical outcome(s) monitored in this study
3. Comparison of baseline rSO2 values (room air and oxygen supplemented) to all collected clinical variables to assess for possibly significant associations
4. Explore the potential impact of rSO2 monitoring on changing the surgical conduct of the procedure Methodology: Single center, prospective, randomized, controlled clinical pilot study Number of Subjects: 100 subjects with balanced randomization (1:1) to control (blinded NIRS data) or intervention (open NIRS data) cohorts Main Criteria for Inclusion: Elderly patients (> 65 years of age) scheduled for a thoracic surgical procedure at UHCMC that will involve SLV.

Duration of Treatment: Cerebral oximetry monitoring will begin with an assessment of both room air and oxygen supplemented bi-frontal baseline NIRS values and continue through the surgery to either PACU discharge or the initial 12 hours of post surgical ICU treatment. Mini Mental Status exam testing and Delirium testing with the Confusion Assessment Method will occur preoperatively and postoperatively through post-operative day (POD) #3 (or discharge if that occurs sooner than POD #3). Enrolled subjects will be followed during the index hospitalization and will undergo a 30 day follow up telephone interview to assess their progress following hospital discharge.

Criteria for Evaluation:

A large number of intraoperative and postoperative clinical variables that include cerebral oximetry, pulse oximetry, blood pressure, a composite outcome measure and clinical variables representing organ function will be assessed with the primary endpoint being the determination of which clinical variables are improved, if any, as a result of being randomized to open NIRS data monitoring with a predefined desaturation intervention algorithm guideline. The Mini Mental Status exam and Confusion Assessment Method test will be used to determine if any measured clinical variables have an effect upon neuropsychological outcomes. The frequency and effectiveness of the various cerebral desaturation mitigating interventions will be assessed in the intervention cohort.

Additional Safety Observations:

The frequency and severity of adverse clinical events and serious adverse clinical events will be assessed to determine if the use of open NIRS data bi-frontal cerebral monitoring is associated with any significant change in the observation of such events.

Statistical Methods:

Preoperative demographics and clinical variables will be compared in the two groups to assess for significant differences using the independent t-test. Differences in the observed clinical data between groups will be determined with the Wilcoxon rank-sum test. Stepwise, forward, multivariable logistic regression analysis will be performed to assess for relationships between cerebral desaturations and any of the measured clinical variables with a p value < 0.05 being considered significant

ELIGIBILITY:
Inclusion Criteria:

1. Any male or female patient ≥ 65 years of age and able to provide informed consent (or consent may be provided by a legally authorized representative) who is scheduled for a thoracic surgical procedure that is expected to involve the use of intraoperative single lung ventilation (SLV)
2. Able to adequately complete a baseline mini-mental status examination (MMSE)
3. Able to complete a baseline confusion assessment method (CAM) examination
4. Able to obtain bi-frontal baseline rSO2 values prior to induction of anesthesia

Exclusion Criteria:

1. Any patient who has participated in a clinical study of an investigational drug or device in the past 30 days
2. Any patient who the principal investigator feels at any time or for any reason should not participate in this clinical study
3. Withdrawal of informed consent for any reason

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 74 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2016-11-10 (Actual); Study Completion 2016-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John C Klick, MD, Principal Investigator — University Hospitals Cleveland Medical Center; Edwin G Avery, MD, Study Director — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Case Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Background] Avery EG. Cerebral oximetry is frequently a "first alert" indicator of adverse outcomes. White paper. October 2010. http://www.somanetics.com/images/stories/pdfs/white-paper-series.pdf Last accessed 08-05-2012
- [Background] Casati A, Fanelli G, Pietropaoli P, Proietti R, Tufano R, Danelli G, Fierro G, De Cosmo G, Servillo G; Collaborative Italian Study Group on Anesthesia in Elderly Patients. Continuous monitoring of cerebral oxygen saturation in elderly patients undergoing major abdominal surgery minimizes brain exposure to potential hypoxia. Anesth Analg. 2005 Sep;101(3):740-747. doi: 10.1213/01.ane.0000166974.96219.cd. PMID 16115985
- [Background] Murkin JM, Adams SJ, Novick RJ, Quantz M, Bainbridge D, Iglesias I, Cleland A, Schaefer B, Irwin B, Fox S. Monitoring brain oxygen saturation during coronary bypass surgery: a randomized, prospective study. Anesth Analg. 2007 Jan;104(1):51-8. doi: 10.1213/01.ane.0000246814.29362.f4. PMID 17179242
- [Background] Tang L, Kazan R, Taddei R, Zaouter C, Cyr S, Hemmerling TM. Reduced cerebral oxygen saturation during thoracic surgery predicts early postoperative cognitive dysfunction. Br J Anaesth. 2012 Apr;108(4):623-9. doi: 10.1093/bja/aer501. Epub 2012 Feb 5. PMID 22311364

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Started | 38 | 36
Completed | 36 | 36
Not Completed | 2 | 0
Not completed — Surgery canceled | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring | Total
Number analyzed (Participants) | 38 | 36 | 74
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 38 | 35 | 73
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 21 | 37
  Male | 22 | 15 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 5 | 3 | 8
  White | 30 | 32 | 62
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: The Primary Objective of This Pilot Study is to Identify the Most Relevant Clinical Outcome Variables Which Significantly Diverge as a Result of Being Randomized to the Intervention Cohort vs. the Control Cohort.
Description: The clinical endpoints are defined by the clinical outcome variables assessed and include relationship of assignment group and AUC of cerebral desats and their observed relationship to PACU/hospital/ICU LOS, AUC of mean arterial blood pressure, IV vasoactive drugs, intraop mLs urine/kg/hr in OR, red blood cell(RBC) transfusion, change in surgical procedure, intra/postop stroke/TIA/MI/afib/AUC glucose > 110 mg/dL, OR time, narcotic administered in the OR, volume of crystalloid/colloid administered in the OR, Anti-emetic meds administered in the OR, Surgical procedure performed, Time on single lung ventilation, Intraop Use of epidural catheter, aldrete PACU score, frequency/severity of N/V in the PACU/ICU, mech vent time in the PACU/ICU, need for postop skilled nursing facility/rehab hospital, need for hospital readmission, change in MMSE/CAM scores from baseline, change in renal fxn compared to baseline, return of bowel function time, postop infection, postop composite endpoint
Time Frame: One year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Relationship of Assignment Group to PACU Length of Stay.
Description: Relationship of assignment group (i.e. control vs intervention group) to PACU LOS
Time Frame: One year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Relationship of Area Under the Curve (AUC) of Cerebral Desaturations to PACU LOS
Description: Relationship of AUC of cerebral desats to PACU LOS
Time Frame: One year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Relationship of Assignment Group to Hospital Length of Stay (HLOS)
Description: Relationship of assignment group (i.e. control vs intervention group) to HLOS
Time Frame: One Year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Relationship of Area Under the Curve (AUC) of Cerebral Desaturations to HLOS
Description: Relationship of Area under the curve (AUC) of cerebral desaturations to HLOS
Time Frame: One year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

6. Primary Outcome: Relationship of Assignment Group to ICU LOS
Description: Relationship of assignment group to ICU LOS
Time Frame: One year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

7. Primary Outcome: Relationship of AUC Cerebral Desaturations to ICU LOS
Description: Relationship of AUC cerebral desaturations to ICU LOS
Time Frame: One year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

8. Primary Outcome: Relationship of Assignment Group to AUC of Mean Arterial Blood Pressure
Description: Relationship of assignment group to AUC of mean arterial blood pressure
Time Frame: One Year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

9. Primary Outcome: Relationship of AUC Cerebral Desaturations to AUC of Mean Arterial Blood Pressure
Description: Relationship of AUC cerebral desaturations to AUC of mean arterial blood pressure
Time Frame: One Year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

10. Primary Outcome: Relationship of AUC Cerebral Desaturations to AUC of Mean Arterial Blood Pressure
Description: Relationship of AUC cerebral desaturations to AUC of mean arterial blood pressure
Time Frame: One year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

11. Primary Outcome: Relationship of AUC Cerebral Desaturations to AUC of Mean Arterial Blood Pressure
Description: Relationship of AUC cerebral desaturations to AUC of mean arterial blood pressure
Time Frame: One year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

12. Primary Outcome: Relationship of Assignment Group to Observed Intraoperative mLs Urine/kg/hr
Description: Relationship of assignment group to observed intraoperative mLs urine/kg/hr
Time Frame: One year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

13. Primary Outcome: Relationship of AUC Cerebral Desaturations to Observed Intraoperative mLs Urine/kg/hr
Description: Relationship of AUC cerebral desaturations to observed intraoperative mLs urine/kg/hr
Time Frame: One year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

14. Primary Outcome: Relationship of Assignment Group to Transfusion of Red Blood Cells
Description: Relationship of assignment group to transfusion of red blood cells
Time Frame: One year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

15. Primary Outcome: Relationship of AUC Cerebral Desaturations to Transfusion of Red Blood Cells
Description: Relationship of AUC cerebral desaturations to transfusion of red blood cells
Time Frame: One year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

16. Primary Outcome: Relationship of Assignment Group to Observed Frequency of Any Change in Surgical Procedure
Description: Relationship of assignment group to observed frequency of any change in surgical procedure
Time Frame: One year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

17. Primary Outcome: Relationship of AUC Cerebral Desaturations to Observed Frequency of Any Change in Surgical Procedure
Description: Relationship of AUC cerebral desaturations to observed frequency of any change in surgical procedure
Time Frame: One year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

18. Primary Outcome: Relationship of Assignment Group to Observed Frequency of Intraoperative or Postoperative Stroke
Description: Relationship of assignment group to observed frequency of intraoperative or postoperative stroke
Time Frame: One Year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

19. Primary Outcome: Relationship of AUC Cerebral Desaturations to Observed Frequency of Intraoperative or Postoperative Stroke
Description: Relationship of AUC cerebral desaturations to observed frequency of intraoperative or postoperative stroke
Time Frame: One year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

20. Primary Outcome: Relationship of Assignment Group to Observed Frequency of Transient Ischemic Attack
Description: Relationship of assignment group to observed frequency of transient ischemic attack
Time Frame: One year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

21. Primary Outcome: Relationship of AUC Cerebral Desaturations to Observed Frequency of Transient Ischemic Attack
Description: Relationship of AUC cerebral desaturations to observed frequency of transient ischemic attack
Time Frame: One year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

22. Primary Outcome: Relationship of Assignment Group to Observed Frequency of Myocardial Infarction
Description: Relationship of assignment group to observed frequency of myocardial infarction
Time Frame: One year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

23. Primary Outcome: Relationship of AUC Cerebral Desaturations to Observed Frequency of Myocardial Infarction
Description: Relationship of AUC cerebral desaturations to observed frequency of myocardial infarction
Time Frame: One year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

24. Primary Outcome: Relationship of Assignment Group to Observed Frequency of Atrial Fibrillation
Description: Relationship of assignment group to observed frequency of atrial fibrillation
Time Frame: One year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

25. Primary Outcome: Relationship of AUC Cerebral Desaturations to Observed Frequency of Atrial Fibrillation
Description: Relationship of AUC cerebral desaturations to observed frequency of atrial fibrillation
Time Frame: One year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

26. Primary Outcome: Relationship of Assignment Group to Observed Frequency of AUC Glucose > 110 mg/dL
Description: Relationship of assignment group to observed frequency of AUC glucose > 110 mg/dL
Time Frame: One year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

27. Primary Outcome: Relationship of AUC Cerebral Desaturations to Observed Frequency of AUC Glucose > 110 mg/dL
Description: Relationship of AUC cerebral desaturations to observed frequency of AUC glucose > 110 mg/dL
Time Frame: One year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

28. Primary Outcome: Relationship of Assignment Group to Observed Operating Room Time
Description: Relationship of assignment group to observed operating room time
Time Frame: One year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

29. Primary Outcome: Relationship of AUC Cerebral Desaturations to Observed Operating Room Time
Description: Relationship of AUC cerebral desaturations to observed operating room time
Time Frame: One year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

30. Primary Outcome: Relationship of Assignment Group to Observed Amount of Narcotic Administered in the Operating Room
Description: Relationship of assignment group to observed amount of narcotic administered in the operating room
Time Frame: One year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

31. Primary Outcome: Relationship of AUC Cerebral Desaturations to Observed Amount of Narcotic Administered in the Operating Room
Description: Relationship of AUC cerebral desaturations to observed amount of narcotic administered in the operating room
Time Frame: One year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

32. Primary Outcome: Relationship of Assignment Group to Observed Volume of Crystalloid/Colloid Administered in the Operating Room
Description: Relationship of assignment group to observed volume of crystalloid/colloid administered in the operating room
Time Frame: One year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

33. Primary Outcome: Relationship of AUC Cerebral Desaturations to Observed Volume of Crystalloid/Colloid Administered in the Operating Room
Description: Relationship of AUC cerebral desaturations to observed volume of crystalloid/colloid administered in the operating room
Time Frame: One year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

34. Primary Outcome: Relationship of Assignment Group to Observed Amount of Anti-emetic Meds Administered in the Operating Room
Description: Relationship of assignment group to observed amount of anti-emetic meds administered in the operating room
Time Frame: One year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

35. Primary Outcome: Relationship of AUC Cerebral Desaturations to Observed Amount of Anti-emetic Meds Administered in the Operating Room
Description: Relationship of AUC cerebral desaturations to observed amount of anti-emetic meds administered in the operating room
Time Frame: One year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

36. Primary Outcome: Relationship of Assignment Group to Reported Surgical Procedure Performed
Description: Relationship of assignment group to reported surgical procedure performed
Time Frame: One year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

37. Primary Outcome: Relationship of AUC Cerebral Desaturations to Reported Surgical Procedure Performed
Description: Relationship of AUC cerebral desaturations to reported surgical procedure
Time Frame: One year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

38. Primary Outcome: Relationship of Assignment Group to Observed Time on Single Lung Ventilation
Description: Relationship of assignment group to observed time on single lung ventilation
Time Frame: One year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

39. Primary Outcome: Relationship of AUC Cerebral Desaturations to Observed Time on Single Lung Ventilation
Description: Relationship of AUC cerebral desaturations to observed time on single lung ventilation
Time Frame: One year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

40. Primary Outcome: Relationship of Assignment Group to Observed Use of Epidural Catheter
Description: Relationship of assignment group to observed use of epidural catheter
Time Frame: One year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

41. Primary Outcome: Relationship of AUC Cerebral Desaturations to Observed Use of Epidural Catheter
Description: Relationship of AUC cerebral desaturations to observed use of epidural catheter
Time Frame: One year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

42. Primary Outcome: Relationship of Assignment Group to Observed Post Anesthesia Care Unit Aldrete Score
Description: Relationship of assignment group to observed post anesthesia care unit Aldrete score
Time Frame: One year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

43. Primary Outcome: Relationship of AUC Cerebral Desaturations to Observed Post Anesthesia Care Unit Aldrete Score
Description: Relationship of AUC cerebral desaturations to observed post anesthesia care unit Aldrete score
Time Frame: One year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

44. Primary Outcome: Relationship of Assignment Group to Observed Frequency and Severity of Nausea/Vomiting in the Post Anesthesia Care Unit/Intensive Care Unit
Description: Relationship of assignment group to observed frequency and severity of nausea/vomiting in the post anesthesia care unit/intensive care unit
Time Frame: One year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

45. Primary Outcome: Relationship of AUC Cerebral Desaturations to Observed Frequency and Severity of Nausea/Vomiting in the Post Anesthesia Care Unit/Intensive Care Unit
Description: Relationship of AUC cerebral desaturations to observed frequency and severity of nausea/vomiting in the post anesthesia care unit/intensive care unit
Time Frame: One year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

46. Primary Outcome: Relationship of Assignment Group to Observed Duration of Mechanical Ventilation in the Post Anesthesia Care Unit/Intensive Care Unit
Description: Relationship of assignment group to observed duration of mechanical ventilation in the post anesthesia care unit/intensive care unit
Time Frame: One year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

47. Primary Outcome: Relationship of AUC Cerebral Desaturations to Observed Duration of Mechanical Ventilation in the Post Anesthesia Care Unit/Intensive Care Unit
Description: Relationship of AUC cerebral desaturations to observed duration of mechanical ventilation in the post anesthesia care unit/intensive care unit
Time Frame: One year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

48. Primary Outcome: Relationship of Assignment Group to Observed Need for Postoperative Discharge to Skilled Nursing/Rehabilitation Facility
Description: Relationship of assignment group to observed need for postoperative discharge to skilled nursing/rehabilitation facility
Time Frame: One year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

49. Primary Outcome: Relationship of AUC Cerebral Desaturations to Observed Need for Postoperative Discharge to Skilled Nursing/Rehabilitation Facility
Description: Relationship of AUC cerebral desaturations to observed need for postoperative discharge to skilled nursing/rehabilitation facility
Time Frame: One year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

50. Primary Outcome: Relationship of Assignment Group to Observed Need for Hospital Readmission
Description: Relationship of assignment group to observed need for hospital readmission
Time Frame: One year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

51. Primary Outcome: Relationship of AUC Cerebral Desaturations to Observed Need for Hospital Readmission
Description: Relationship of AUC cerebral desaturations to observed need for hospital readmission
Time Frame: One year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

52. Primary Outcome: Relationship of Assignment Group to Observed Change in CAM or MMSE Scores From Baseline
Description: Relationship of assignment group to observed change in CAM or MMSE scores from baseline
Time Frame: One year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

53. Primary Outcome: Relationship of AUC Cerebral Desaturations to Observed Change in CAM or MMSE Scores From Baseline
Description: Relationship of AUC cerebral desaturations to observed change in CAM or MMSE scores from baseline
Time Frame: One year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

54. Primary Outcome: Relationship of Assignment Group to Observed Change in Renal Function From Baseline
Description: Relationship of assignment group to observed change in renal function from baseline
Time Frame: One year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

55. Primary Outcome: Relationship of AUC Cerebral Desaturations to Observed Change in Renal Function From Baseline
Description: Relationship of AUC cerebral desaturations to observed change in renal function from baseline
Time Frame: One year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

56. Primary Outcome: Relationship of Assignment Group to Observed Time to Return of Bowel Function Time
Description: Relationship of assignment group to observed time to return of bowel function time
Time Frame: One year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

57. Primary Outcome: Relationship of AUC Cerebral Desaturations to Observed Time to Return of Bowel Function Time
Description: Relationship of AUC cerebral desaturations to observed time to return of bowel function time
Time Frame: One year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

58. Primary Outcome: Relationship of Group Assignment to Any Observed Postoperative Infection
Description: Relationship of group assignment to any observed postoperative infection
Time Frame: One year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

59. Primary Outcome: Relationship of AUC Cerebral Desaturations to Any Observed Postoperative Infection
Description: Relationship of AUC cerebral desaturations to any observed postoperative infection
Time Frame: One year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

60. Primary Outcome: Relationship of Assignment Group to Observed Time to Wean From Postoperative Supplemental Oxygen
Description: Relationship of assignment group to observed time to wean from postoperative supplemental oxygen
Time Frame: One year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

61. Primary Outcome: Relationship of AUC Cerebral Desaturations to Observed Time to Wean From Postoperative Supplemental Oxygen
Description: Relationship of AUC cerebral desaturations to observed time to wean from postoperative supplemental oxygen
Time Frame: One year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

62. Primary Outcome: Relationship of Assignment Group to Observed Incidence of Postop Morbidity Composite Endpoint (Defined in Description Section Below)
Description: Relationship of assignment group to observed incidence of postop morbidity composite endpoint (defined by having any 1 of the following: new onset afib, ≥Grade 2 PONV, HLOS≥4.5 days, PACU LOS≥2 hours, any infection, death, stroke, MI, greater 0.5 mg/dL increase in Cr or new need for renal dialysis, postop need for IV inotropes or vasoactive meds)
Time Frame: One year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

63. Primary Outcome: Relationship of AUC Cerebral Desaturations to Observed Incidence of Postoperative Morbidity Composite Endpoint (Defined in Description Section Below)
Description: Relationship of AUC cerebral desaturations to observed incidence of postoperative morbidity composite endpoint (defined by having any one of the following: new onset atrial fibrillation, ≥Grade 2 PONV, HLOS≥4.5 days, PACU LOS≥2 hours, any infectious complication, death, stroke, myocardial infarction, greater 0.5 mg/dL increase in creatinine or new need for renal dialysis, postoperative need for intravenous inotropes or vasoactive medications)
Time Frame: One year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

64. Secondary Outcome: Assess the Frequency of Cerebral Desaturations in Both Cohorts by Examining Both the Total Number of Patients Experiencing Any Cerebral Desaturation as Well as the Total Number of Events Among Patients Experiencing Any Cerebral Desaturation.
Description: Assess the frequency of cerebral desaturations in both the intervention and control cohorts by examining both the total number of patients experiencing any cerebral desaturation as well as the total number of events among patients experiencing any cerebral desaturation.
Time Frame: one year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

65. Secondary Outcome: Adverse Clinical Events and Serious Adverse Events Overall and in Each Cohort
Description: Assess the frequency of adverse clinical events and serious adverse events overall and in each cohort
Time Frame: one year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

66. Secondary Outcome: Perform a Comprehensive Assessment of the Frequency and Efficacy of Predefined rSO2 Desaturation Mitigation Interventions and Their Collective Ability to Affect the Observed Cerebral Oximetry Values.
Description: Perform a comprehensive assessment of the frequency and efficacy of predefined rSO2 desaturation mitigation interventions (e.g., increase MAP with IV vasoconstrictor or fluid bolus, normalize ETCO2, deepen anesthesia, etc.) and their collective ability to affect the observed cerebral oximetry values. This will allow determination of the average number of interventions required and those most commonly effective in mitigating desaturation.
Time Frame: one year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

67. Secondary Outcome: Assess the Interventional Cohort's Preoperative Demographics and Collected Covariates for Association With the Ease or Difficulty of Mitigating Observed Cerebral Desaturation Events.
Description: Because mitigating cerebral desaturations involves increasing oxygen delivery to the tissue it is possible that there is a relationship between preoperative demographic/variables such as age, peripheral vascular disease, left ventricular dysfunction, COPD, etc. and the ability to effectively mitigate desaturations in that subjects with disease in these organ systems may be more resistant to responding to desaturation interventions.
Time Frame: one year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

68. Other Pre Specified Outcome: • Logistic Regression Analysis to Determine the Most Relevant AUCrSO2 Desaturation Value(s) Associated With Any Detrimental Clinical Outcome(s) Monitored in This Study
Description: Logistic regression analysis to determine the most relevant AUCrSO2 desaturation value(s) associated with any detrimental clinical outcome(s) monitored in this study
Time Frame: one year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

69. Other Pre Specified Outcome: Logistic Regression Analysis to Determine the Most Relevant AUC Blood Pressure Values Associated With Any Detrimental Clinical Outcome(s) Monitored in This Study
Description: Logistic regression analysis to determine the most relevant AUC blood pressure values associated with any detrimental clinical outcome(s) monitored in this study
Time Frame: one year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

70. Other Pre Specified Outcome: Comparison of Baseline rSO2 Values (Room Air and Oxygen Supplemented) to All Collected Clinical Variables to Assess for Possibly Significant Associations
Description: Comparison of baseline rSO2 values (room air and oxygen supplemented) to all collected clinical variables to assess for possibly significant associations
Time Frame: One year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

71. Other Pre Specified Outcome: Explore the Potential Impact of rSO2 Monitoring on Changing the Surgical Conduct of the Procedure
Description: Explore the potential impact of rSO2 monitoring on changing the surgical conduct of the procedure
Time Frame: one year
Population: Data not collected
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Not collected
Description: Adverse events data was not collected.
Arm/Group | Intervention Cohort | Blinded Cerebral Oximetry Monitoring
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-04): https://cdn.clinicaltrials.gov/large-docs/57/NCT01866657/Prot_SAP_000.pdf